CLINICAL TRIAL: NCT01277263
Title: Predicting Pathological Response Within the 1st Week of Neoadjuvant Chemotherapy Using Functional Parameters Measured With Diffuse Optical Spectroscopic Imaging
Brief Title: Predicting Pathological Response Within the 1st Week of Chemotherapy Using Diffuse Optical Spectroscopic Imaging
Status: Withdrawn | Type: Observational
Why Stopped: Not a Clinical Trial study
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg, PhD., Director, Beckman Laser Institute and Medical Clinic, Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20107789
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — C-Protein serum
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy Imaging — Monitoring Breast Cancer during chemo therapy

SUMMARY:
Women with Breast Cancer who do not respond to chemotherapy may undergo months of treatment with little or no change in tumor size or overall outcome.

The Researchers have demonstrated a previously undescribed "metabolic flare" response observed very early in neoadjuvant treatment in breast cancer patients. The research can determine that this flare is predictive of overall therapy response and is due to both an inflammatory reaction and cell death induced by cytotoxic therapy.

DETAILED DESCRIPTION:
The researcher can use Diffuse Optical Spectroscopic Imaging device to measure and predict the markers of the response in the first weeks of chemo-therapy.

The oxyhemoglobin flare response can predictive of overall pathological response to chemotherapy in human subjects. These vascular changes can indicate the rapid transient increase and then decrease in oxyhemoglobin concentration in the first hours and days after therapeutic administration. The magnitude and time course of the flare response in patients receiving cytotoxic therapy will differ between pathological responders and non-responders. This oxyhemoglobin "flare response" can be observed In tumors where vascular dynamics are intact.

ELIGIBILITY:
Inclusion Criteria:

* Female, not pregnant, not breastfeeding
* greater than 21 years of age but less than 75 years of age
* will be receiving neoadjuvant chemotherapy for breast cancer as prescribed by their oncologist

Exclusion Criteria:

* Under 21 year of age
* Female pregnant or breastfeeding

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from an outpatient population of the Cancer Center Clinic, Beckman Laser Medical Clinic of University of California, Irvine and UCI Pacific Breast Care. Subjects with the requisite diagnosis of breast cancer will be candidates for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
improve treatment prognosis for breast cancer patients | 12 weeks
  The proposed research plan has the ability to significantly impact breast cancer research and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tromberg, PhD, Study Director — Beckman Laser Institute
Locations (3):
- United States (3):
  - Pacific Breast Care Medical Clinic, Costa Mesa, California
  - Beckman Laser Institute, Irvine, California
  - Chao Family Comprehensive Cancer Center, UCIMC, Orange, California